CLINICAL TRIAL: NCT00109369
Title: Vermont Diabetes Information System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Vermont Program for Quality in Health Care (Other)
Responsible Party: Benjamin Littenberg, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61167 (completed); R01DK061167 (NIH); K24DK068380 (NIH)
Record Dates: First submitted 2005-04-27; First posted 2005-04-27 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus
Keywords: Chronic Disease; Multi-Hospital Information Systems; Clinical Decision Support Systems; Reminder Systems; Registries; Quality of Healthcare; Guideline Adherence; Outcome and Process Assessment (Health Care); Technology Assessment, Biomedical; Primary Health Care; Hypercholesterolemia; Hypertension; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Chronic Disease; Hypercholesterolemia; Hypertension; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Provider and patient receive Diabetes Information System services
  Interventions: Other: Information and decision support for providers and patients
- Control (No Intervention): Usual Care

INTERVENTIONS:
Other: Information and decision support for providers and patients — Laboratory-based decision support, reminders, and population report cards.
  Other Names: Vermedx Diabetes Information System
  Arms: Active

SUMMARY:
The Vermont Diabetes Information System (VDIS) is a registry-based decision support and reminder system based on the Chronic Care Model and targeted to primary care physicians and their patients with diabetes. It will be evaluated by a randomized, controlled study in 60 Primary Care practices in Vermont and nearby New York.

DETAILED DESCRIPTION:
The long-term goal of the Vermont Diabetes Information System is to reduce morbidity and mortality from diabetes mellitus. The project will implement and evaluate a state-wide system to support evidence-based disease management by primary care providers, their practices, and their patients in the community. The primary study question is: "What is the effect of a Diabetes Information System (including education, feedback and decision support) upon disease control measured by glycated hemoglobin?" Secondary questions address the effect of the system upon adherence to guideline recommendations, blood pressure control, patient satisfaction, medication use, and functional status. We hypothesize that the information system will result in improvements in the process and outcomes of clinical care. There are two specific aims:

Aim 1: Implement the Diabetes Information System. Objective 1.1: Develop a registry of patients with diabetes in primary care practices in Vermont; Objective 1.2: Provide education and feedback to providers regarding their patients with diabetes; Objective 1.3: Deliver decision support (flow sheets, alerts and reminders) based on the registry and targeted at primary care providers and patients, to prompt ideal management of diabetes.

Aim 2: Assess the Diabetes Information System. Objective 2.1: Assess disease control and guideline adherence by examining registry data in all subjects in a prospective, two-year, randomized, controlled trial in 60 primary care practices; Objective 2.2: Assess outcomes (blood pressure control, obesity, functional status, symptoms, medication use, and satisfaction) by interview and examination in a sub-sample of patients from the controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Diabetes confirmed by Primary Care provider

Exclusion Criteria:

* Severe dementia
* Nursing home resident

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7500 (Estimated)
Dates: Start 2003-06; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 2 years

SECONDARY OUTCOMES:
Processes of care | 2 years
Blood pressure control | 2 years
Hypercholesterolemia | 2 years
Adherence to Practice Guidelines | 2 years
Quality of life | 2 years
Healthcare utilization | 2 years
Patient satisfaction | 2 years
Medication use | 2 years
Functional status | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Littenberg, MD, Principal Investigator — University of Vermont; Charles D. MacLean, MDCM, Study Director — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

REFERENCES:
- [Background] MacLean CD, Littenberg B, Gagnon M, Reardon M, Turner PD, Jordan C. The Vermont Diabetes Information System (VDIS): study design and subject recruitment for a cluster randomized trial of a decision support system in a regional sample of primary care practices. Clin Trials. 2004;1(6):532-44. doi: 10.1191/1740774504cn051oa. PMID 16279294